CLINICAL TRIAL: NCT03658252
Title: A Randomised Controlled Trial Assessing the Efficacy of Targeted Intervention for Topical Steroid Phobia.
Brief Title: Efficacy of Targeted Intervention for Topical Steroid Phobia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Health System, Singapore (Other)
Responsible Party: Principal Investigator, Ellie Choi, Senior Resident, Division of Dermatology, Department of Medicine, Principal Investigator, National University Health System, Singapore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2018/00481
Record Dates: First submitted 2018-08-31; First posted 2018-09-05 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Dermatologic Disease; Phobia; Adherence, Medication
Keywords: steroid phobia; topical corticosteroids; eczema; psoriasis; adherence; quality of life
MeSH Terms: conditions — Skin Diseases; Phobic Disorders; Medication Adherence; Eczema; Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in the intervention arm will be shown a 2 minute educational video, and given an information leaflet on topical steroids. At 1 month of follow up, a link encouraging participants to sign up for a pre-selected, disease specific, moderated online support group would be sent to their emails.
  Participants will continue to receive standard medical care and counselling by their dermatologists as clinically indicated.
  Interventions: Behavioral: Targeted education; Behavioral: Online disease specific forum
- Control (No Intervention): Patients in the control arm will receive only standard medical care and counseling by their dermatologist as clinically indicated.

INTERVENTIONS:
Behavioral: Targeted education — Educational video developed by the hospital, addressing common misconceptions of topical steroids. A patient information leaflet on topical steroids
  Arms: Intervention
Behavioral: Online disease specific forum — An invitation to join an online moderated disease specific social forum
  Arms: Intervention

SUMMARY:
Topical steroids are an important component of treatment for many dermatological conditions, however 'Corticosteroid phobia' is a significant factor contributing to non adherence to prescribed therapy.

The primary aim of this study is to determine the effectiveness of targeted education, and involvement in a moderated social forum in reducing steroid phobia as assessed by the TOPICOP© score. Secondary objectives include determining if a decrease in TOPICOP© score correlates to an increase in compliance, or an improvement in quality of life.

DETAILED DESCRIPTION:
Oral and topical steroids are commonly prescribed in the dermatological setting for its anti inflammatory property, for conditions ranging from eczematous disease, autoimmune disorders and many other primary dermatoses.

There is large evidence that topical steroids are safe in the long term when used appropriately, and the benefits of reducing skin inflammation outweigh their risks of skin atrophy and telangiectasia.

Topical corticosteroid phobia (TCS phobia) toward topical steroids is a significant factor contributing to non adherence. Much of this may be attributed to the excessive or exaggerated propagation of 'steroid phobia' messages from the internet, family/friends, and even medical professionals.

The TOPICOP© score is the first, and presently only score that is validated to explore TCS phobia. It consists of 12 items assessing three domains of TCS phobia, knowledge and beliefs, fears and behavior. Responses are graded with a 4 point Likert scale.

The primary aim of this study is to determine the effectiveness of targeted education, and involvement in a moderated social forum in reducing steroid phobia as assessed by the TOPICOP© score. Secondary objectives include determining if reduction in steroid phobia correlates to an increase in compliance, or an improvement in quality of life.

The investigators hypothesise that providing information directed at common misconceptions towards topical steroids will decrease steroid phobia, and that this would result in improved adherence and quality of life. Providing access to moderated forums with balanced views and information may also help to address concerns of patients.

ELIGIBILITY:
Inclusion Criteria:

Participants aged 21 years and above. Currently prescribed and expected to be on topical steroids for the next 3 months.

Willing to provide telephone number or email address, and to be recontacted. Able to read and understand english.

Exclusion Criteria:

Not on topical steroids. Unable to understand english. Unable or unwilling to be contacted for follow up surveys.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-05-04 (Actual)

PRIMARY OUTCOMES:
Change in TOPICOP© score at 3 months | 3 months
  Validated score assessing topical corticosteroid (TCS) phobia. It consists of 12 items assessing three domains of TCS phobia, knowledge and beliefs, fears and behaviour on a 4 point likert scale. The individual domain and global scores are calculated as a percentage of the total score. A higher score indicated greater steroid phobia.

SECONDARY OUTCOMES:
Change in TOPICOP© score at 1 month | 1 month
  Validated score assessing topical corticosteroid (TCS) phobia. It consists of 12 items assessing three domains of TCS phobia, knowledge and beliefs, fears and behaviour on a 4 point likert scale. The individual domain and global scores are calculated as a percentage of the total score. A higher score indicated greater steroid phobia.
Change in ECOB (Elaboration d'un outil d'evaluation de l'observance des traitements médicamenteux) score at 1 month | 1 month
  Score comprising 4 questions to assess patients awareness of their medication and compliance. Questions administered in english. Designed initially to assess adherence to topical and oral therapies in acne, but is used in this study to assess adherence to topical steroids. Range of total score is from 0-4. A score of 4 classifies the patient as adherent, and <4 as non adherent.
Change in ECOB (Elaboration d'un outil d'evaluation de l'observance des traitements médicamenteux) score at 3 month | 3 month
  Score comprising 4 questions to assess patients awareness of their medication and compliance. Questions administered in english. Designed initially to assess adherence to topical and oral therapies in acne, but is used in this study to assess adherence to topical steroids. Range of total score is from 0-4. A score of 4 classifies the patient as adherent, and <4 as non adherent.
Change in Dermatology Life Quality Index score at 1 month | 1 month
  Dermatology specific quality of life instrument. A 10 point questionnaire, with a total score range from 0 to 30. A higher score indicated greater impact on quality of life.
Change in Dermatology Life Quality Index score at 3 month | 3 month
  Dermatology specific quality of life instrument. A 10 point questionnaire, with a total score range from 0 to 30. A higher score indicated greater impact on quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ellie Choi, MBBS, MRCP, MMed (IM), Principal Investigator — National University Healthcare System; Chris Tan, MBBS, FAMS, Study Director — National University Healthcare System; Nisha Chandran, MBBS, MRCP, MMed (IM), Study Director — National University Healthcare System
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pawin H, Beylot C, Chivot M, Faure M, Poli F, Revuz J, Dreno B. Creation of a tool to assess adherence to treatments for acne. Dermatology. 2009;218(1):26-32. doi: 10.1159/000165628. Epub 2008 Oct 22. PMID 18946201
- [Background] Dreno B, Thiboutot D, Gollnick H, Finlay AY, Layton A, Leyden JJ, Leutenegger E, Perez M; Global Alliance to Improve Outcomes in Acne. Large-scale worldwide observational study of adherence with acne therapy. Int J Dermatol. 2010 Apr;49(4):448-56. doi: 10.1111/j.1365-4632.2010.04416.x. PMID 20465705
- [Background] Moret L, Anthoine E, Aubert-Wastiaux H, Le Rhun A, Leux C, Mazereeuw-Hautier J, Stalder JF, Barbarot S. TOPICOP(c): a new scale evaluating topical corticosteroid phobia among atopic dermatitis outpatients and their parents. PLoS One. 2013 Oct 16;8(10):e76493. doi: 10.1371/journal.pone.0076493. eCollection 2013. PMID 24146878